CLINICAL TRIAL: NCT05330533
Title: Effect of Recent Ejaculation on Scrotal Duplex Parameters in Infertile Males With Varicocele
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Thabet Mohamed Ali Elsebaity, Principal investigator , resident doctor, Assiut University
Other Study IDs: Ejaculation effect on Duplex
Record Dates: First submitted 2022-03-16; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-03

CONDITIONS: Varicocele
MeSH Terms: conditions — Varicocele

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: scrotal duplex — Scrotal colour doppler ultrasonography

SUMMARY:
Evaluate the effect of recent ejaculation on scrotal duplex parameters in infertile males with varicocele

DETAILED DESCRIPTION:
Varicocele is abnormal dilatation of the pampiniform plexus veins draining the testicles.

It manifests as an abnormal retrograde flow in the internal spermatic venous system or dilation of venous branches in the external cremasteric system .

It affects approximately 15% in the general population, 35 - 40% in men with primary infertility and approximately 80% of men with secondary infertility. It could often concomitantly occur with infertility or chronic scrotal pain causing impaired spermatogenesis and is the most common correctable cause of male infertility. it may affects spermatogenesis via different mechanisms such as increased testicular heat, hormonal disorders and reflux of toxic metabolites.

Scrotal colour Doppler ultrasonography (USG) is a widely used method for evaluation of varicocele patients . It can be used along with physical examination in these patients through evaluation of vein reflux and diameter; in cases where palpation may be problematic. Furthermore, the degree of reflux and vein diameter can be used during the decision-making stage while treating varicocele .

Ejaculation is the process by which sperms move from epididymis via vas deferens to urethra and finally expelled out through the urethral meatus by the contraction of smooth muscles. A normal antegrade ejaculation consists of emission, expulsion (ejection), and orgasm .

In the evaluation of infertile patients, semen analysis is required for evaluation of number, motility and morphology of spermatozoa with scrotal colour Doppler USG. Ejaculation for the purpose of sperm analysis is known to significantly increase testicular blood supply .

ELIGIBILITY:
Inclusion Criteria:

1. Infertile male patients.
2. patients with scrotal varicocele.
3. male patients aging over 18 years old.

Exclusion Criteria:

1. Pyospermia.
2. Epididymitis.
3. Orchitis.
4. Anejaculation.
5. Recurrent varicocele.
6. Patients who previously underwent scrotal or inguinal surgery.

Ages: 18 Years to 65 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Effect of Recent( Ejaculation) on Scrotal Duplex Parameters in Infertile( Males) With Varicocele
Study Population: Infertile male patients with scrotal varicocele aging over 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of varicose vein diameter pre and post ejaculation. | within 30 minutes post ejaculation
  Assessment of the change in varicose vein diameter by scrotal colour doppler ultrasonography pre ejaculation and within 30 minutes post ejaculation.

SECONDARY OUTCOMES:
Assessment of varicose vein reflux time pre and post ejaculation. | Within 30 minutes post ejaculation
  Assessment of varicose vein reflux time by scrotal duplex pre ejaculation and within 30 minutes post ejaculation.

REFERENCES:
- [Background] Kizilkan Y, Duran MB, Senel S, Yikilmaz TN, Akbelen B, Toksoz S. The effect of ejaculation time on varicose vein diameter and reflux level. Andrologia. 2021 Aug;53(7):e14090. doi: 10.1111/and.14090. Epub 2021 Apr 28. PMID 33913191
- [Background] Bello JO, Bhatti KH, Gherabi N, Philipraj J, Narayan Y, Tsampoukas G, Shaikh N, Papatsoris A, Moussa M, Buchholz N. The usefulness of elastography in the evaluation and management of adult men with varicocele: A systematic review. Arab J Urol. 2021 Sep 16;19(3):255-263. doi: 10.1080/2090598X.2021.1964256. eCollection 2021. PMID 34552777
- [Background] Senturk AB, Cakiroglu B, Yaytokgil M, Aydin C, Sungur M, Akkoc A. Effect of venous reflux time on testosterone and semen parameters of infertile males after microscopic varicocelectomy. Andrologia. 2020 Jul;52(6):e13583. doi: 10.1111/and.13583. Epub 2020 Apr 9. PMID 32271466
- [Background] Sihag P, Tandon A, Pal R, Jain BK, Bhatt S, Kaur S, Sinha A. Sonography in male infertility: a look beyond the obvious. J Ultrasound. 2018 Sep;21(3):265-276. doi: 10.1007/s40477-018-0294-5. Epub 2018 Mar 28. PMID 29594932
- [Background] Raveendran AV, Agarwal A. Premature ejaculation - current concepts in the management: A narrative review. Int J Reprod Biomed. 2021 Jan 25;19(1):5-22. doi: 10.18502/ijrm.v19i1.8176. eCollection 2021 Jan. PMID 33553999